CLINICAL TRIAL: NCT06628713
Title: On Demand Treatment of Angioedema Attacks in Adolescent and Adult Post-Trial and Naive Patients 12 Years and Older With Hereditary Angioedema (HAE) Type I or II With Sebetralstat
Brief Title: Treatment of Angioedema Attacks in Adolescent and Adult Patients 12 Years and Older With HAE Type I or II With Sebetralstat
Status: Approved for marketing | Type: Expanded Access
Sponsor: KalVista Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: KVD900-EAP-US-1
Record Dates: First submitted 2024-09-26; First posted 2024-10-08 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Hereditary Angioedema
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — sebetralstat

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Sebetralstat — Oral Plasma Kallikrein Inhibator
  Other Names: KVD900

SUMMARY:
The sebetralstat Early Access Program (EAP) provides early access to the investigational medicinal product (IMP) sebetralstat to eligible and approved Type I or II Hereditary Angioedema (HAE) adolescent and adult post-trial and naïve patients for the on-demand treatment of angioedema attacks where the treating Physician determines they might benefit from this treatment.

ELIGIBILITY:
Inclusion Criteria:

* At least 12 years of age.
* Able to provide written, informed consent or assent.
* Confirmed diagnosis of HAE Type I or II.

Exclusion Criteria:

* Confirmed diagnosis of HAE with nC1-INH or acquired angioedema.
* Confirmed pregnancy or breast-feeding.
* Any clinically significant medical condition or medical history that, in the opinion of the Treating Physician, would interfere with the patient's safety.
* Known hypersensitivity to sebetralstat or its excipients.
* Patient with a medical history or known to have severe hepatic impairment (Child Pugh C).
* Patients who require sustained use of strong cytochrome P450 3A4 inhibitors or inducers.

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- KalVista Investigative Site, Scottsdale, Arizona, United States